CLINICAL TRIAL: NCT07201025
Title: Imaging Assessments of ARPKD Kidney Disease Progression
Acronym: IMAGE-ARPKD
Status: Recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Katherine Dell, Professor of Pediatrics, The Cleveland Clinic
Other Study IDs: 24-088; 2R01DK114425 (NIH)
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Autosomal Recessive Polycystic Kidney Disease
Keywords: MRI; ARPKD; Pediatric; Ciliopathy; Biomarker
MeSH Terms: conditions — Polycystic Kidney, Autosomal Recessive; Ciliopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Early CKD Patients: eGFR > or = to 90 ml/min/1.73m2
- Mild CKD Patients: eGFR 60-89 ml/min/1.73m2
- Moderate CKD Patients: eGFR 30-59 ml/min/1.73m2
- Healthy Controls

SUMMARY:
Autosomal Recessive Polycystic Kidney Disease (ARPKD) is a potentially lethal genetic disorder for which there are currently no disease specific treatments. Clinical trials have been limited by the absence of robust measures of disease progression. The overall goal of this 5 year NIH-funded prospective, observational multicenter study conducted at CC (primary site) and Children's Hospital of Philadelphia (CHOP) (collaborating site) is establish a set of rapid, quantitative, and reproducible novel kidney MRI measures applicable to standard clinical MRI scanners, which could serve as potential biomarkers to measure response to therapy in patients across the disease spectrum and all ages.

The investigators will recruit a total of 45 ARPKD patients and 15 healthy controls at the the two sites . All subjects will be > or = 6yrs old with no contraindications to undergoing MRI (non contrast). ARPKD subjects will be recruited into one of 3 cohorts based on their estimated glomerular filtration rate (eGFR): early CKD (eGFR> or =90ml/min/1.73m2), mild CKD (60-89ml/min/1.73m2) and moderate CKD (30-59ml/min/1.73m2). For ARPKD subjects, participation will last 3 years and consist of a baseline and 3 subsequent annual visits. Healthy controls will only have 1 study visit. Study visits for all participants will include collection of clinical and demographic data, clinical blood and urine tests (E.g. serum creatinine) and MRI imaging. ARPKD (but not healthy subjects) will also undergo a measured GFR test (iohexol clearance) to accurately assess their kidney function.

DETAILED DESCRIPTION:
Autosomal Recessive Polycystic Kidney Disease (ARPKD) is a potentially lethal genetic disorder that affects approximately 1/20,000 children and shares common cellular pathophysiology with other cystic kidney diseases, including Autosomal Dominant PKD (ADPKD). The genetics, pathology and clinical features of ARPKD, however, are distinct from ADPKD. In ARPKD, diffuse fusiform dilatations of the collecting tubules ("microcysts") predominate rather than the macrocysts seen in ADPKD. ARPKD kidneys may be very large at presentation, but, unlike ADPKD, actually stabilize in size as normal parenchyma is replaced by cysts and progressive fibrosis develops. ARPKD morbidity and mortality is significant: 30% of children die as neonates and 40-50% of survivors progress to end-stage kidney disease (ESKD) by age 18. Importantly, there are currently no disease-specific, clinically-available therapies for ARPKD and treatment is limited to chronic kidney disease (CKD) management. Several novel therapies have shown promise in ARPKD animal models. Unfortunately, there are currently no reliable clinical measures of ARPKD progression that show changes over a several year period of a clinical trial except in the most severely affected young children, creating a roadblock for implementing clinical trials for ARPKD therapies, especially in patients with less advanced disease.

Conventional endpoints for CKD progression, e.g., 50% decline in estimated glomerular filtration rate (eGFR) or progression to ESKD have substantial limitations in assessing ARPKD progression. Studies from 2 prospective observational cohorts found that the rates of GFR decline in ARPKD patients was relatively slow but also highly variable. Magnetic Resonance Imaging (MRI) measures of total kidney volume (TKV), which have been used successfully in ADPKD trials, are generally not applicable to ARPKD, since TKV does not increase with progressive disease except in severely affected young patients. Therefore, there is a critical need for new, sensitive biomarkers to enable effective clinical trials of therapies for ARPKD. Quantitative MRI techniques, including novel Magnetic Resonance Fingerprinting (MRF), Arterial Spin Labelling (ASL) and Magnetic Resonance Elastography (MRE), have the potential to provide measurable assessments of kidney structure and function. The overall objective of this multi-site study is to establish a set of rapid, quantitative, and reproducible kidney MRI methods applicable to standard clinical MRI scanners, which could serve as potential biomarkers to risk stratify ARPKD patients for clinical trial enrollment and measure response to therapy across the kidney disease spectrum and all ages.

The Aims of this study are (1) to determine the capability of multimodal MRI biomarkers to accurately and repeatably detect and stage ARPKD kidney disease across the full spectrum of disease from early-stage CKD characterized by diffuse kidney cysts (MRF) and reduced kidney perfusion (ASL) to later-stage CKD characterized by progressive kidney fibrosis (MR elastography, MRE); (2) to determine the sensitivity of these MRI biomarkers to detect changes in ARPKD kidney disease progression over time in comparison to gold-standard GFR assessments; and (3) to determine the feasibility of a new free-breathing MRF methodology that would allow infants and young children to be scanned without sedation. For these studies, the investigators will recruit ARPKD patients ≥6 years of age with early, mild, and moderate CKD from across the US for 4 annual multimodal MRI scans and GFR measurements at two collaborating sites (CC/CWRU and CHOP). Age-matched healthy controls will also be recruited for an MRI scan. If successful, the proposed studies will support use of these multimodal MRI biomarkers as outcome measures and/or high-risk subject enrichment for future clinical trials for ARPKD patients.

ELIGIBILITY:
Inclusion criteria:

ALL SUBJECTS

* Ages >6 years old
* Able to lay still for 30 minutes in an MRI scanner ARPKD Patients
* Clinical and/or genetic diagnosis of ARPKD
* eGFR (creatinine based) >30ml/min/1.732 performed within the last year Healthy Controls
* Otherwise healthy with no known structural or functional kidney disease
* No history of hypertension or documented high blood pressure within the last year

Exclusion criteria:

ALL SUBJECTS

* Contraindications to MRI (e.g. metal implants)
* Parental/patient refusal to sign an informed consent/ assent form ARPKD Patients
* Prior kidney or other solid organ transplant
* eGFR <30ml/min/1.732 Healthy Controls
* Systemic diseases known to place patient at risk for kidney disease (e.g. diabetes mellitus)
* Obesity (BMI >95th percentile for age for <18 years old, or BMI>30 for adults)
* History of prematurity (<32 weeks gestational age)

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Inclusion criteria:
  ALL SUBJECTS
  * Ages >6 years old
  * Able to lay still for 30 minutes in an MRI scanner ARPKD Patients
  * Clinical and/or genetic diagnosis of ARPKD
  * eGFR >30ml/min/1.732 performed within the last year Healthy Controls
  * Otherwise healthy with no known structural or functional kidney disease
  * Normal documented blood pressure within the last year
  Exclusion criteria:
  ALL SUBJECTS
  * Contraindications to MRI (e.g. metal implants)
  * Parental/patient refusal to sign an informed consent/ assent form ARPKD Patients
  * Prior kidney or other solid organ transplant
  * eGFR <30ml/min/1.732 and/or anticipated dialysis or kidney transplant within the next 3 years Healthy Controls
  * Systemic diseases known to place patient at risk for kidney disease (e.g. diabetes mellitus)
  * Obesity (BMI >95th percentile for age for <18 years old, or BMI>30 for adults)
  * History of prematurity (<32 weeks)
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2029-02-28 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
The diagnostic performance (AUROC, sensitivity, specificity) of the multimodal MRI assessments MRF (mean kidney T1 and T2), ASL (mean kidney perfusion), and MRE (mean kidney stiffness), alone or in combination to differentiate the 4 study cohorts | 3 Years
The relationship between the imaging biomarkers, MRF (mean kidney T1 and T2), ASL (mean kidney perfusion), and MRE (mean kidney stiffness) alone or in combination, to baseline and change in measured GFR over 3 years in the 3 ARPKD cohorts | 3 Years
The level of agreement between breath-hold and free breathing kidney MRF assessments in the 4 cohorts | 3 Years

SECONDARY OUTCOMES:
Repeatability of multimodal MRI assessments in ARPKD and healthy control subjects | 3 years
Reproducibility of findings at the two study sites | 3 Years

CONTACTS AND LOCATIONS:
Overall Officials: Katherine M Dell, MD, Principal Investigator — The Cleveland Clinic
Locations (2):
- United States (2):
  - Cleveland Clinic, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] MacAskill CJ, Kretzler ME, Parsons A, Gange V, Hach J, Larson S, Zhu Y, Perino J, Farr S, Markley M, Pritts N, Perera-Gonzalez M, Clark HA, Kuehn B, Liu KC, Yu X, Ma D, Chen Y, Flask CA, Dell KM. Multimodal Magnetic Resonance Imaging Assessments of Kidney Disease Severity in Autosomal Recessive Polycystic Kidney Disease. Kidney Int Rep. 2024 Sep 12;9(12):3592-3595. doi: 10.1016/j.ekir.2024.09.006. eCollection 2024 Dec. No abstract available. PMID 39698366
- [Background] MacAskill CJ, Markley M, Farr S, Parsons A, Perino JR, McBennett K, Kutney K, Drumm ML, Pritts N, Griswold MA, Ma D, Dell KM, Flask CA, Chen Y. Rapid B1-Insensitive MR Fingerprinting for Quantitative Kidney Imaging. Radiology. 2021 Aug;300(2):380-387. doi: 10.1148/radiol.2021202302. Epub 2021 Jun 8. PMID 34100680
- [Background] MacAskill CJ, Erokwu BO, Markley M, Parsons A, Farr S, Zhang Y, Tran U, Chen Y, Anderson CE, Serai S, Hartung EA, Wessely O, Ma D, Dell KM, Flask CA. Multi-parametric MRI of kidney disease progression for autosomal recessive polycystic kidney disease: mouse model and initial patient results. Pediatr Res. 2021 Jan;89(1):157-162. doi: 10.1038/s41390-020-0883-9. Epub 2020 Apr 13. PMID 32283547